CLINICAL TRIAL: NCT05239923
Title: COVID19 Oral Vaccine Consisting of Bacillus Subtilis Spores Expressing and Displaying the Receptor Binding Domain of Spike Protein of SARS-COV2
Brief Title: COVID19 Oral Vaccine Consisting of Bacillus Subtilis Spores
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: DreamTec Research Limited (Industry)
Collaborators: Middle East Cell and Gene Therapy (Unknown); National Institute of Genetic Engineering and Biotechnology (Unknown)
Responsible Party: Principal Investigator, Keith Kwong, Chief Scientific Officer, DreamTec Research Limited
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: PRP/008/21FXMiddleEast
Record Dates: First submitted 2022-02-11; First posted 2022-02-15 (Actual); Last update posted 2022-02-15 (Actual); Status verified 2022-02

CONDITIONS: COVID-19 Pneumonia
Keywords: COVID-19; Vaccine Reaction; Bacillus subtilis
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: People were not vaccinated with SARS-COV2 vaccine were recruited for the administration of Bacillus subtilis oral vaccine
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- generation of neutralizing antibody for unvaccinated participants (Experimental): participants received vaccine 1 capsule of 1×10^10 CFU of B. subtilis spore at day 0, 14, and 28 respectively.
  Interventions: Biological: Bacillus subtilis

INTERVENTIONS:
Biological: Bacillus subtilis — Bacillus subtilis, a harmless intestinal commensal, has earned in recent years, great reputation as a vaccine production host and delivery vector with advantages such as low cost, safe for human consumption and straightforward administration. The technology team has succeeded engineering Bacillus subtilis with spore coat proteins resembling the proteins of the nucleus and spikes of coronal virus. This product could have a vaccine like activity within the intestinal environment.

SUMMARY:
This is a study trial to assess the effectiveness of the immune response stimulated by the genetically engineered Bacillus subtilis which express and display Spike protein of the SARS-COV2 on the spore coat.

DETAILED DESCRIPTION:
Bacillus subtilis is regarded as safe organism by The Food and Drug Administration and it is presented in most food sources. Preliminary experiments have shown that the genetically engineered Bacillus subtilis can express and display receptor binding domain of spike protein of the SARS-COV2 on its spore coat, thus successfully inducing the secretion of cytokines of human cells in vitro. Previous experiments also successfully demonstrated that a increased detection of neutralizing IgG and IgM levels in mice and human after oral administrated with the Bacillus subtilis. This suggests that the transgenic spores of Bacillus subtilis have successfully activated the immune system, producing high-affinity neutralizing antibodies and memory B cells. Furthermore, no adverse effects were shown in all the mices. The engineered Bacillus subtilis will be further studied in a human trial through oral administration to test its safety and the immune effect resulted in human bodys.

ELIGIBILITY:
Inclusion Criteria:

* healthy
* age over 12 years
* the outcome of the following examinations should be clinically insignificant: medical and surgical history (hypo-, hypertension, allergy, other diseases, major surgery, micturition, defecation, sleep, illness within the last 4 weeks prior to the start of the trial);
* participant vaccinated with COVID-19 over 6 months
* anti-SARS CoV 2 neutralizing antibody is negative in serum.

Exclusion Criteria:

* pregnant women
* history of COVID-19 infection or showing COVID-19 infection symptoms
* having had contact to people with known COVID-19 infection in the last 14 days
* having fever (> 37.4oC in the last 24 hours), dry cough or feeling tired and having aches and pains, nasal congestion, runny nose, sore throat and diarrhea.

positive real time RT-PCR COVID-19 test.

* persons with autoimmune diseases
* allergic diathesis or any clinically significant allergic disease (i.e. asthma)
* any condition that might impair the immune response
* recent or current immunosuppressive medication
* any other vaccine application 5 months before the first dose

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2021-08-28 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
Safety of the engineered Bacillus subtilis | 3 months
  To measure the blood pressure and number of incidence of adverse event from the beginning of the administration to 30 days after the last administration (3 months)
Concentration of Neutralizing IgG antibody against Receptor binding domain of spike protein of SARS-CoV2 | 2 months
  To measure the concentration of Neutralizing IgG antibody against Receptor binding domain of spike protein of SARS-CoV2 before the administration and 14, 28 days after the administration (2 month)

CONTACTS AND LOCATIONS:
Locations (2):
- DreamTec Research Limited, Hong Kong, Hong Kong
- Middle East Cell and Gene Therapy, Tehran, Iran

IPD SHARING:
Plan to Share IPD: No